CLINICAL TRIAL: NCT06308510
Title: Detection of Aneuploidy in Cell Free DNA to Improve the Sensitivity of Diagnostic Peritoneal Lavage in Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. B. (Bianca) Mostert, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2024 0533
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer
Keywords: peritoneal metastasis; cfDNA
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peritoneal lavage fluid, which may contain cfDNA in non-cancer controls and gastric cancer patients, and blood in gastric cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Gastric cancer patients: Operable patients who will undergo DLS for GC. Patients will be identified from the MDT (multidisciplinary tumor board).
  Interventions: Other: collection additional peritoneal lavage fluid
- non-cancer controls: Patients who will undergo a planned laparoscopy for bariatric or gallbladder disease
  Interventions: Other: collection additional peritoneal lavage fluid

INTERVENTIONS:
Other: collection additional peritoneal lavage fluid — collection additional peritoneal lavage fluid

SUMMARY:
Aneuploidy may be used as a more sensitive diagnostic tool to detect peritoneal metastasis compared to conventional cytology and imaging techniques. Our aim is to establish whether aneuploidy as detected in cfDNA (as a measure for ctDNA) in PLF of patients with GC may hold value as an additional staging and tumor evaluation method in GC patients.

DETAILED DESCRIPTION:
To ensure the appropriate treatment strategy for gastric cancer, various methods are employed to determine clinical disease stage. Peritoneal metastases are common in gastric cancer, but accurately detecting these peritoneal metastasis using conventional imaging techniques remains challenging. To increase the sensitivity of staging when gastric cancer appears resectable on CT imaging, a diagnostic peritoneal staging laparoscopy (DLS) is performed. During DLS, the abdominal cavity is inspected for the presence of macroscopic peritoneal metastasis. Furthermore, a peritoneal lavage with saline is performed, and the collected fluid is examined by a pathologist for the presence of cancer cells. However, the sensitivity of this cytological evaluation is limited, and as a result of false negative results, patients currently unjustly undergo treatment with curative intent, exposing them to the risks and side-effects of surgery and intensive perioperative chemotherapy. A more sensitive technique to detect peritoneal metastases during staging would lead to better personalized treatment; less toxic palliative treatment, or more intensive peritoneum-directed therapy in a trial setting in selected patients.

A more sensitive diagnostic tool to detect peritoneal metastasis compared to conventional cytology and imaging techniques may be the detection of ctDNA. One way to detect ctDNA is by assessing aneuploidy, as its presence reflects the fraction of circulating tumor DNA within cell-free DNA.

Objective:To assess the value of ctDNA detection using aneuploidy analyses of peritoneal lavage fluid using mFAST-SeqS method in a prospective cohort of patients with gastric cancer who undergo a staging laparoscopy, in addition to the current staging methods (cytology, radiology, laparoscopy) and blood ctDNA analysis.

ELIGIBILITY:
Gastric cancer patients:

Inclusion Criteria:

* Age ≥18 years old;
* Written informed consent according to the ICH-GCP and national/local regula-tions.

Exclusion Criteria:

- Language difficulty, dementia or altered mental status prohibiting the under-standing and giving of informed consent.

non-cancer controls:

Inclusion criteria:

* Operable patients who will undergo a planned diagnostic laparoscopy for a benign indication bariatric or gallbladder disease);
* Age ≥18 years old;
* Written informed consent according to the ICH-GCP and national/local regulations.

Exclusion criteria:

* Active inflammation or infection;
* Subjects with previous malignancies are excluded unless a complete remission was achieved at least 5 years prior to study entry (exceptions include but are not limited to, non-melanoma skin cancers; in situ bladder cancer, or in situ co-lon cancers; in situ cervical cancers/dysplasia; or breast carcinoma in situ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients:
  Patients who will undergo DLS for GC or GEJ carcinoma
  Non-cancer controls:
  Operable patients who will undergo a planned diagnostic laparoscopy for a benign indication (bariatric or gallbladder disease);
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity mFast-SeqS | 4 years
  The primary endpoint is the sensitivity of the mFast-SeqS technique in patients with GC, and refers to the ability of the mFast-SeqS technique to correctly identify patients with the pres-ence of tumor cells in the peritoneal cavity.

SECONDARY OUTCOMES:
DFS | 2 years
  No locoregional or distant recurrence of disease,
Concordance detection rates peritoneal dissemination | 4 years
  • Concordance of detection rates of peritoneal dissemination will be analyzed using cohen's kappa/mcNemar's test

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Mostert, MD, Principal Investigator — Erasmus Medical Center; Sjoerd Lagarde, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No